CLINICAL TRIAL: NCT00582712
Title: An Initial Study of Lithium in Patients With Medullary Thyroid Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Budget/Funding
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CO07312; 2007-0195 (Other: Institutional Review Board); NCI-2011-00714 (Registry Identifier: NCI Trial ID)
Record Dates: First submitted 2007-12-19; First posted 2007-12-28 (Estimated); Results first posted 2016-12-12 (Estimated); Last update posted 2019-12-09 (Actual); Status verified 2016-10

CONDITIONS: Medullary Thyroid Cancer
Keywords: medullary thyroid cancer; lithium
MeSH Terms: conditions — Carcinoma, Medullary | interventions — Lithium Carbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lithium Capsules (Experimental): Lithium carbonate
  Interventions: Drug: Lithium carbonate

INTERVENTIONS:
Drug: Lithium carbonate — Lithium 300mg by mouth, three times daily, escalating to a lithium level of 0.8-1.2; Continue until progressive disease/unacceptable toxicity; Evaluate every 4 weeks.

SUMMARY:
Primary objective is to evaluate the tumor response rate of patients with MTC treated with Lithium carbonate

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed MTC with signs of residual/persistent disease based on tumor marker levels and/or radiographic imaging. Pathologic diagnosis must be confirmed at UWCCC. Grading must be confirmed by pathologic review performed at UWCCC.
* Elevated neuroendocrine markers at least 1 month post -op. In MTC, persistently elevated neuroendocrine markers such as calcitonin and CEA are indicative of persistent disease.
* Disease progression is not required for this trial

  * 4 weeks from the completion of major surgery, chemotherapy, or other systemic therapy or local liver therapy to study registration. Subjects will have had standard of care prior to enrollment. Subjects will have had standard of care prior to enrollment (for example it could include total thyroidectomy, central lymph node dissection, and when necessary ipsilateral radical neck dissection but is tailored to the patient).
  * 3 weeks from the completion of radiation therapy to study registration
* The following laboratory values obtained within 14 days prior to registration:

  * Absolute neutrophils count (ANC) ≥ 1000/mm3
  * Platelets ≥ 75,000/mm3
  * Hemoglobin ≥ 8.0 g/dL
  * Total bilirubin greater than or equal to 2.0 X the upper limit of normal (ULN)
  * AST greater than or equal to 3 X ULN or greater than or equal to 5 X ULN if liver metastases are present
  * Creatinine greater than or equal to ULN
  * Serum sodium within normal limits
* ECOG performance status of 2
* Capable of understanding the investigational nature, potential risks and benefits of the study, and able to provide valid informed consent.
* Availability of tissue specimens to be analyzed for pathologic confirmation.
* Age ≥ 18 years.
* Women must not be pregnant or lactating due to the deleterious effects of Lithium carbonate on a fetus or small child. All females of childbearing potential must have a blood test or urine study within 2 weeks prior to registration to rule out pregnancy.
* Women of childbearing potential and sexually active males are required to use an accepted and effective method of contraception.
* Patients must not have known history of allergic reactions or adverse reactions to Lithium or its derivatives.
* Patients are not allowed to be on concurrent chemotherapy or radiation therapy.

Exclusion Criteria:

* Gastrointestinal tract disease resulting in an inability to take oral medication (i.e. ulcerative disease, uncontrolled nausea, vomiting, diarrhea, bowel obstruction, or inability to swallow the tablets).
* Significant, active cardiac disease
* Patients must not be taking the following medications: diuretics, ACE inhibitors, NSAIDs (except aspirin or sulindac), neuroleptics, tetracycline, and COX2 inhibitors.
* Patients with radiographic evidence of disease will be presented the option to undergo a tumor biopsy although this is not mandatory.
* Patients already taking Lithium for any reason are not allowed on study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2008-01; Primary Completion 2009-05 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herbert Chen, MD, Principal Investigator — University of Wisconsin Cancer Center
Locations (1):
- Uniersity of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin, United States

REFERENCES:
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study recruited participants from a large cancer research institution in Wisconsin from December 2007 through May 2008.
Groups:
- Lithium Capsules: Lithium carbonate: Lithium 300mg by mouth, three times daily, escalated to a lithium level of 0.8-1.2; Continued until progressive disease/unacceptable toxicity; Evaluated every 4 weeks.
Period: Overall Study
Arm/Group | Lithium Capsules
Started | 5
Completed | 1
Not Completed | 4
Not completed — Adverse Event | 1
Not completed — Lack of Efficacy | 1
Not completed — Withdrawal by Subject | 1
Not completed — Complicating disease requiring treatment | 1

BASELINE CHARACTERISTICS:
Population: This study enrolled participants with Medullary Thyroid Cancer (MTC).
Arm/Group | Lithium Capsules
Number analyzed (Participants) | 5
Age, Customized [Number; unit: participants]
  < 50 years of age | 1
  50-59 years of age | 2
  60-69 years of age | 1
  > 69 years of age | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response Rate Measured by the Response Evaluation Criteria in Solid Tumors (RECIST)
Time Frame: 1 year
Population: No data was ever analyzed, resulted, or published on this study.
Arm/Group | Lithium Capsules
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected starting on of after Day 0 up to 4 years.
Description: Adverse events (AEs) were reported routinely at scheduled times during the trial. Additionally, some adverse events were reported in an expedited manner for more timely monitoring of patient safety and care. The serum lithium level was checked after 4-5 days of treatment by blood sample prior to daily dose 1 of lithium. If lithium level was outside the 0.8-1.2 mmol/L range, lithium levels were monitored weekly for 4 weeks and monthly after 4 weeks.
  AEs grades range from 1 (mild) to 5 (death).
Arm/Group | Lithium Capsules
Serious Adverse Events (participants affected / at risk) | 4/5
Other Adverse Events (participants affected / at risk) | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lithium Capsules (N=5)
Death (General disorders) | 3 (3) — Death not associated with CTCAE term - Death was unrelated to study.
Grade 3 fatigue (General disorders) | 1 (1)
Grade 3 speech impairment (Nervous system disorders) | 1 (1)
Grade 2 dizziness (vertigo) (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No